CLINICAL TRIAL: NCT03002792
Title: Neurodevelopment Outcomes After Pediatric Dental Caries Treatment Under General Anaesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Hui Zhang, M.D., Ph.D. Director and Professor, Department of Anaesthesiology, School of Stomatology, Air Force Military Medical University, China
Other Study IDs: 2014KTCL03_05
Record Dates: First submitted 2016-12-17; First posted 2016-12-26 (Estimated); Last update posted 2017-11-28 (Actual); Status verified 2017-01

CONDITIONS: Anesthesia
Keywords: anesthesia; neurodevelopment; dental caries
MeSH Terms: conditions — Dental Caries | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- general anesthesia: caries treatment under general anesthesia
  Interventions: Procedure: general anesthesia
- caries treatment only: caries treatment without general anesthesia

INTERVENTIONS:
Procedure: general anesthesia — nitrous oxide, sevoflurane, propofol, cisatracurium, fentanyl for induction and maintenance with sevoflurane
  Groups: general anesthesia

SUMMARY:
The purpose of this study is to investigate whether early expose to general anaesthesia will influence neurodevelopment.

DETAILED DESCRIPTION:
Participants, according to the state of illness and clinical requirements, assigned to receive dental caries treatment with or without general anesthesia. During the follow-up, various of neurodevelopment assessment will be done at specific timepoint to investigate whether general anaesthesia will influence neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age>=36 weeks
* American Society of Anesthesiologists（ASA） physical status Ⅰ or Ⅱ，with very limited systemic disease.
* Age<=6 yr

Exclusion Criteria:

* did not provide research authorization；
* unable to contact or inconvenient for follow-up;
* hypersensitive to general anesthesia drug;
* previous exposure to general anesthesia in utero;
* previous exposure to general anesthesia as a neonate
* previous exposure to psychotropic medication;
* complications at birth such as low weigh, hypoxia, or cerebral edema;
* any other known diseases may influence the neurodevelopment

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients revieve carves treatment in Department of Pediatric Dentistry，School of Stomatology, the Fourth Military Medical University
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Full Scale Intelligence Quotient (IQ) | 24-28 weeks after enrollment
  according to Wechsler Preschool and Primary Scale of Intelligence fourth edition (WPPSI-IV)

SECONDARY OUTCOMES:
Verbal Comprehension Index | 24-28 weeks after enrollment
  according to WPPSI-IV
Visual Spatial Index | 24-28 weeks after enrollment
  according to WPPSI-IV
Fluid Spatial Index | 24-28 weeks after enrollment
  according to WPPSI-IV
Working Memory Index | 24-28 weeks after enrollment
  according to WPPSI-IV
Processing Speed Index | 24-28 weeks after enrollment
  according to WPPSI-IV
Executive Function | 24-28 weeks after enrollment
  according to Behavior Rating Inventory of Executive Function-Preschool Version (BRIEF-P)
Adaptive Behavior | 24-28 weeks after enrollment
  according to Adaptive Behavior Assessment System second edition
Emotion Comprehension | 24-28 weeks after enrollment
  according to Test of Emotion Comprehension(TEC) (designed by Pons & Harris ,2000)

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhang, M.D., Study Director — School of Stomatology, the Fourth Military Medical University
Locations (1):
- School of Stomatology, the Fourth Military Medical University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zou X, Liu F, Zhang X, Patterson TA, Callicott R, Liu S, Hanig JP, Paule MG, Slikker W Jr, Wang C. Inhalation anesthetic-induced neuronal damage in the developing rhesus monkey. Neurotoxicol Teratol. 2011 Sep-Oct;33(5):592-7. doi: 10.1016/j.ntt.2011.06.003. Epub 2011 Jun 25. PMID 21708249
- [Background] Paule MG, Li M, Allen RR, Liu F, Zou X, Hotchkiss C, Hanig JP, Patterson TA, Slikker W Jr, Wang C. Ketamine anesthesia during the first week of life can cause long-lasting cognitive deficits in rhesus monkeys. Neurotoxicol Teratol. 2011 Mar-Apr;33(2):220-30. doi: 10.1016/j.ntt.2011.01.001. Epub 2011 Jan 15. PMID 21241795
- [Background] Shen X, Liu Y, Xu S, Zhao Q, Guo X, Shen R, Wang F. Early life exposure to sevoflurane impairs adulthood spatial memory in the rat. Neurotoxicology. 2013 Dec;39:45-56. doi: 10.1016/j.neuro.2013.08.007. Epub 2013 Aug 27. PMID 23994303
- [Background] Hansen TG, Pedersen JK, Henneberg SW, Pedersen DA, Murray JC, Morton NS, Christensen K. Academic performance in adolescence after inguinal hernia repair in infancy: a nationwide cohort study. Anesthesiology. 2011 May;114(5):1076-85. doi: 10.1097/ALN.0b013e31820e77a0. PMID 21368654
- [Background] Ing C, DiMaggio C, Whitehouse A, Hegarty MK, Brady J, von Ungern-Sternberg BS, Davidson A, Wood AJ, Li G, Sun LS. Long-term differences in language and cognitive function after childhood exposure to anesthesia. Pediatrics. 2012 Sep;130(3):e476-85. doi: 10.1542/peds.2011-3822. Epub 2012 Aug 20. PMID 22908104
- [Background] Wilder RT, Flick RP, Sprung J, Katusic SK, Barbaresi WJ, Mickelson C, Gleich SJ, Schroeder DR, Weaver AL, Warner DO. Early exposure to anesthesia and learning disabilities in a population-based birth cohort. Anesthesiology. 2009 Apr;110(4):796-804. doi: 10.1097/01.anes.0000344728.34332.5d. PMID 19293700
- [Background] Graham MR, Brownell M, Chateau DG, Dragan RD, Burchill C, Fransoo RR. Neurodevelopmental Assessment in Kindergarten in Children Exposed to General Anesthesia before the Age of 4 Years: A Retrospective Matched Cohort Study. Anesthesiology. 2016 Oct;125(4):667-677. doi: 10.1097/ALN.0000000000001245. PMID 27655179
- [Background] Sun LS, Li G, Miller TL, Salorio C, Byrne MW, Bellinger DC, Ing C, Park R, Radcliffe J, Hays SR, DiMaggio CJ, Cooper TJ, Rauh V, Maxwell LG, Youn A, McGowan FX. Association Between a Single General Anesthesia Exposure Before Age 36 Months and Neurocognitive Outcomes in Later Childhood. JAMA. 2016 Jun 7;315(21):2312-20. doi: 10.1001/jama.2016.6967. PMID 27272582
- [Background] Davidson AJ, Disma N, de Graaff JC, Withington DE, Dorris L, Bell G, Stargatt R, Bellinger DC, Schuster T, Arnup SJ, Hardy P, Hunt RW, Takagi MJ, Giribaldi G, Hartmann PL, Salvo I, Morton NS, von Ungern Sternberg BS, Locatelli BG, Wilton N, Lynn A, Thomas JJ, Polaner D, Bagshaw O, Szmuk P, Absalom AR, Frawley G, Berde C, Ormond GD, Marmor J, McCann ME; GAS consortium. Neurodevelopmental outcome at 2 years of age after general anaesthesia and awake-regional anaesthesia in infancy (GAS): an international multicentre, randomised controlled trial. Lancet. 2016 Jan 16;387(10015):239-50. doi: 10.1016/S0140-6736(15)00608-X. Epub 2015 Nov 4. PMID 26507180